CLINICAL TRIAL: NCT02425111
Title: An Open-Label Phase 3b Study to Assess Mucosal Healing in Subjects With Moderately to Severely Active Crohn's Disease Treated With Vedolizumab IV
Brief Title: Effect of Intravenous (IV) Vedolizumab on Mucosal Healing in Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLN0002-3028; U1111-1159-5806 (Registry Identifier: WHO); 2014-003509-13 (EudraCT Number); 183974 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2015-03-26; First posted 2015-04-23 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vedolizumab 300 mg (Experimental): Part A: Vedolizumab 300 mg, intravenously (IV), once on Day 1 and Weeks 2, 6, 14 and 22, followed by Part B: Vedolizumab 300 mg, intravenously (IV), once at Weeks 30, 38, and 46.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous injection
  Other Names: MLN0002

SUMMARY:
The purpose of this study is to evaluate endoscopic remission at Week 26 as assessed by ileocolonoscopy.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have Crohn's disease. This study will look at mucosal healing in people who take vedolizumab.

The study will enroll approximately 100 patients and will be conducted in 2 Parts. Part A will consist of a 26-week treatment period and all participants will receive vedolizumab 300 mg intravenously (IV) on Day 1 and at Weeks 2, 6, 14 and 22. Part B will consist of a 26-week extension treatment period and all participants will receive vedolizumab 300 mg IV at Weeks 30, 38, and 46.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 70 weeks for Parts A, B and 18-Week Follow-up combined. Participants will make multiple visits to the clinic. All participants included in the study will also have a 6 month safety follow-up telephone call following his/her last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a diagnosis of moderately to severely active Crohn's disease (CD) at least 3 months prior to enrollment, with a Crohn's Disease Activity Index (CDAI) score of 220-450 during the Screening Period, a simple endoscopic score for Crohn's Disease (SES-CD) score of ≥7 and presence of at least one mucosal ulceration documented by recorded ileocolonoscopy at Screening assessed by the central reader.
4. Has CD with involvement of the ileum and/or colon that can be assessed by ileocolonoscopy.
5. Is male or female and aged 18 to 80 years, inclusive.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 18 weeks after last dose.
8. Has demonstrated an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents as defined below:

   * Immunomodulators:

     i. Has signs and symptoms of persistently active disease despite a history of at least one 12-week regimen of oral azathioprine (≥1.5 mg/kg) or 6-mercaptopurine (≥0.75 mg/kg), OR ii. Has a history of intolerance (including but not limited to nausea/vomiting, abdominal pain, pancreatitis, liver function test abnormalities, lymphopenia, thiopurine S-methyltransferase non wild type [where wild type is defined as thiopurine S-methyltransferase (TPMT)*1/*1], infection) to at least 1 immunomodulator.
   * Tumor necrosis factor- alpha (TNF-α) antagonists:

     i. Has signs and symptoms of persistently active disease despite a history of at least 1 induction with:
     1. Infliximab: 4-week regimen of 5 mg/kg, 2 doses at 2 weeks apart, OR
     2. Adalimumab: 2-week regimen of 160 mg on Day 1 and 80 mg on Day 15, OR
     3. Certolizumab: 4-week regimen of 400 mg initially at Weeks 0, 2, 4 OR ii. Has recurrence of symptoms during maintenance dosing following prior clinical benefit (discontinuation despite clinical benefit does not qualify), OR iii. Has a history of intolerance of infliximab, adalimumab, or certolizumab, including but not limited to, infusion-related reaction, demyelination, congestive heart failure, or infection.
   * Corticosteroids i. Signs and symptoms of persistently active disease despite a history of at least one 4-week induction regimen that included a dose equivalent to prednisone 30 mg daily orally for 2 weeks or intravenous(ly) (IV) for 1 week, OR ii. Signs and symptoms of persistently active disease despite treatment with budesonide 9 mg daily or 6 mg daily for maintenance, OR iii. At least one failed attempt to taper corticosteroids to below a dose equivalent to prednisone 10 mg daily orally, OR iv. History of intolerance to corticosteroids (including, but not limited to, Cushing's syndrome, osteopenia/osteoporosis, hyperglycemia, insomnia, and infection).
9. May be receiving a stable therapeutic dose of conventional therapies for CD (excluding other biologic agents 60 days before enrollment).
10. Has a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factors must be up-to-date on colorectal cancer surveillance (may be performed during Screening).

Exclusion Criteria:

1. Has received a diagnosis of ulcerative colitis or indeterminate colitis.
2. Has clinical evidence of abdominal abscess.
3. Has a history of >3 small bowel resections or diagnosis of short bowel syndrome.
4. Has extensive colonic resection, ie, subtotal or total colectomy with <15 cm colon remaining.
5. Has ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
6. Has a history or evidence of adenomatous colonic polyps that have not been removed.
7. Has a history or evidence of colonic mucosal dysplasia.
8. Has intolerance or contraindication to undergo ileocolonoscopy.
9. Has active or latent tuberculosis, regardless of treatment history, as evidenced by any of the following:

   a. History of tuberculosis (TB). b. A diagnostic TB test performed during screening that is positive, as defined by: i. A positive QuantiFERON® test or 2 successive indeterminate QuantiFERON tests OR ii. A tuberculin skin test reaction ≥10 mm (≥5 mm in participants receiving the equivalent of >15 mg/day prednisone).
10. Has chronic hepatitis B (HBV) or hepatitis C (HCV) infection.
11. Has any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
12. Has evidence of active C. difficile infection or is having treatment for C. difficile infection or other intestinal pathogens during Screening.
13. Has evidence of an active infection during Screening.
14. Currently requires or has a planned surgical intervention for CD during the study.
15. Has received any investigational compound within 60 days of enrollment.
16. Has received any biologics within 60 days of enrollment.
17. Has received any live vaccinations within 30 days prior to enrollment.
18. Has conditions which, in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
19. Has any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal (GI), genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.
20. Has a history of hypersensitivity or allergies to vedolizumab or its components.
21. Has had prior exposure to vedolizumab, natalizumab, efalizumab, or rituximab.
22. Had a surgical procedure requiring general anesthesia within 30 days prior to screening or is planning to undergo major surgery during the study period.
23. Has a history of malignancy, except for the following: adequately-treated nonmetastatic basal cell skin cancer; squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to Screening; and history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to screening. Participants with a remote history of malignancy (eg, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to enrollment.
24. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
25. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist during Screening or prior to the administration of study drug.
26. Has any of the following laboratory abnormalities during the Screening Period:

    i. Hemoglobin level <8 g/dL. ii. White blood cell (WBC) count <3*10^9/L. iii. Lymphocyte count <0.5*10^9/L. iv. Platelet count <100*10^9/L or >1200*10^9/L. v. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3*the upper limit of normal (ULN).

    vi. Alkaline phosphatase >3*ULN. vii. Serum creatinine >2*ULN.
27. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to enrollment.
28. Has an active psychiatric problem that, in the investigator's opinion, may interfere with compliance with study procedures.
29. Is unable to attend all the study visits or comply with study procedures.
30. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 18 weeks after participating in this study; or intending to donate ova during such time period.
31. If male, the participant intends to donate sperm during the course of this study or for 18 weeks thereafter.
32. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
33. Participants who are at sites participating in the magnetic resonance enterography (MREn) substudy may not participate if they have intolerance or contraindication to the procedure or if any of the following exclusions apply:

    1. Has certain implanted medical devices, such as pacemakers or implantable cardioverter defibrillators (ICDs), or ferromagnetic metallic foreign bodies, such as shrapnel or certain tattoos.
    2. Has allergy to gadolinium-based magnetic resonance (MR) IV contrast agents.
    3. Has known claustrophobia.
    4. Has estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 at Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2018-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (79):
- United States (22):
  - La Jolla, California
  - Hamden, Connecticut
  - Gainesville, Florida
  - Inverness, Florida
  - Maitland, Florida
  - Miami, Florida
  - Winter Park, Florida
  - Macon, Georgia
  - Suwanee, Georgia
  - Topeka, Kansas
  - Baton Rouge, Louisiana
  - Columbia, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Manhasset, New York
  - Poughkeepsie, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Germantown, Tennessee
- Belgium (6):
  - Bonheiden
  - Brussels
  - Herentals
  - Kortrijk
  - Leuven
  - Roeselare
- Canada (5):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Vaughan, Ontario
- Czechia (4):
  - Hradec Králové
  - Kladno
  - Pardubice
  - Prague
- France (12):
  - Nice, Alpes Maritimes
  - Pessac, Gironde
  - Reims, Marne
  - Lille, Nord
  - Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Lille
  - Nantes
  - Nice
  - Pessac
  - Reims
  - Saint-Etienne
  - Toulouse
- Hungary (14):
  - Békéscsaba
  - Budapest
  - Debrecen
  - Gyöngyös
  - Gyula
  - Jászberény
  - Kistarcsa
  - Miskolc
  - Mosonmagyaróvár
  - Pécs
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Vác
- Italy (11):
  - San Giovanni Rotondo, Foggia
  - Rozzano, Milano
  - San Donato Milanese, Milano
  - Bologna
  - Florence
  - Napoli
  - Padua
  - Roma
  - Rozzano
  - San Donato Milanese
  - San Giovanni Rotondo
- Poland (5):
  - Bialystok
  - Elblag
  - Poznan
  - Warsaw
  - Wroclaw

REFERENCES:
- [Derived] Rimola J, Colombel JF, Bressler B, Adsul S, Siegelman J, Cole PE, Lindner D, Danese S. Magnetic Resonance Enterography Assessment of Transmural Healing with Vedolizumab in Moderate to Severe Crohn's Disease: Feasibility in the VERSIFY Phase 3 Clinical Trial. Clin Exp Gastroenterol. 2024 Jan 27;17:9-23. doi: 10.2147/CEG.S429039. eCollection 2024. PMID 38298861
- [Derived] Narula N, Wong ECL, Dulai PS, Marshall JK, Jairath V, Reinisch W. Comparative Effectiveness of Biologics for Endoscopic Healing of the Ileum and Colon in Crohn's Disease. Am J Gastroenterol. 2022 Jul 1;117(7):1106-1117. doi: 10.14309/ajg.0000000000001795. Epub 2022 Apr 15. PMID 35435862
- [Derived] Danese S, Sandborn WJ, Colombel JF, Vermeire S, Glover SC, Rimola J, Siegelman J, Jones S, Bornstein JD, Feagan BG. Endoscopic, Radiologic, and Histologic Healing With Vedolizumab in Patients With Active Crohn's Disease. Gastroenterology. 2019 Oct;157(4):1007-1018.e7. doi: 10.1053/j.gastro.2019.06.038. Epub 2019 Jul 4. PMID 31279871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 42 investigative sites in Belgium, Canada, Czech Republic, France, Hungary, Italy, Poland and the United States from 30 March 2015 to 21 February 2018.
Pre-assignment Details: Participants with a diagnosis of Crohn's Disease were enrolled and received vedolizumab.
Period: Part A: Treatment Period
Arm/Group | Vedolizumab 300 mg
Started | 101
Completed (Completed=Completed Study Drug) | 78
Not Completed | 23
Not completed — Pretreatment Event/Adverse Event | 2
Not completed — Lack of Efficacy | 15
Not completed — Voluntary Withdrawal | 4
Not completed — Lost to Follow-up | 2
Period: Part B: Treatment Extension Period
Arm/Group | Vedolizumab 300 mg
Started | 56
Completed | 46
Not Completed | 10
Not completed — Pretreatment Event/Adverse Event(s) | 3
Not completed — Lack of Efficacy | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  years | 38.0 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants
    Female | 49
    Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was collected only in the United States. Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants
    Hispanic or Latino | 1
    Non-Hispanic and Latino | 32
    Not Collected | 68
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants
    Asian | 2
    Black or African American | 1
    White | 98
Region of Enrollment [Count of Participants; unit: Participants] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants
    Belgium | 8
    Canada | 14
    Czech Republic | 14
    France | 2
    Hungary | 14
    Italy | 9
    Poland | 7
    United States | 33
Height [Mean (Standard Deviation); unit: cm] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  cm | 172.5 (9.81)
Weight [Mean (Standard Deviation); unit: kg] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  kg | 73.94 (18.795)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  kg/m^2 | 24.71 (5.365)
Smoking Classification [Count of Participants; unit: Participants] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants
    Participant has never smoked | 46
    Participant is a current smoker | 33
    Participant is an ex-smoker | 22
Female Reproductive Status [Count of Participants; unit: Participants] — Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants
    Postmenopausal | 6
    Surgically Sterile | 9
    Female of Childbearing Potential | 34
    N/A (Participant is a Male) | 52
Number of Participants with Endoscopic Remission [Count of Participants; unit: Participants] — Endoscopic remission is defined as a simple endoscopic score for Crohn's Disease (SES-CD) score of ≤4. Population: FAS included all enrolled participants who received at least 1 dose of study drug.
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Achieving Endoscopic Remission at Week 26
Description: Endoscopic remission is defined as a simple endoscopic score for Crohn's Disease (SES-CD) score of ≤4. The SES-CD evaluates 4 endoscopic variables (ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis in 5 segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable is the sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Week 26
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 11.9 [6.3 to 19.8]

2. Secondary Outcome: Part A: Percentage of Participants Achieving Complete Mucosal Healing at Week 26
Description: Complete mucosal healing is defined as absence of ulceration.
Time Frame: Week 26
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 14.9 [8.6 to 23.3]

3. Secondary Outcome: Part B: Percentage of Participants Achieving Complete Mucosal Healing at Week 52
Description: Complete mucosal healing is defined as absence of ulceration.
Time Frame: Week 52
Population: FAS-Extension is the subset of participants in the FAS who were able to be consented for Part B, based on the timing of Amendment 4. FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 56
percentage of participants | 17.9 [8.9 to 30.4]

4. Secondary Outcome: Part A: Percentage of Participants Achieving Endoscopic Remission at Week 14
Description: Endoscopic remission is defined as a SES-CD score of ≤4. The SES-CD evaluates 4 endoscopic variables (ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis in 5 segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable is the sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Week 14
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 16.8 [10.1 to 25.6]

5. Secondary Outcome: Part B: Percentage of Participants Achieving Endoscopic Remission at Week 52
Description: as for outcome 4
Time Frame: Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 56
percentage of participants | 16.1 [7.6 to 28.3]

6. Secondary Outcome: Part A: Percentage of Participants With Endoscopic Response at Week 14
Description: Endoscopic response is defined as a reduction in SES-CD from Baseline by ≥50%. The SES-CD evaluates 4 endoscopic variables (ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis in 5 segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable is the sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Baseline and Week 14
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 33.7 [24.6 to 43.8]

7. Secondary Outcome: Part A: Percentage of Participants With Endoscopic Response at Week 26
Description: as for outcome 6
Time Frame: Baseline and Week 26
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 24.8 [16.7 to 34.3]

8. Secondary Outcome: Part B: Percentage of Participants With Endoscopic Response at Week 52
Description: as for outcome 6
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 56
percentage of participants | 51.8 [38.0 to 65.3]

9. Secondary Outcome: Part A: Percentage of Participants Achieving Clinical Response at Week 10
Description: Clinical response is defined as Crohn's Disease Activity Index (CDAI) decrease from Baseline of ≥100 points. CDAI is a scoring system for the assessment of Crohn's Disease Activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Time Frame: Baseline and Week 10
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 54.5 [44.2 to 64.4]

10. Secondary Outcome: Part A: Percentage of Participants Achieving Clinical Response at Week 26
Description: Clinical response is defined as CDAI decrease from Baseline of ≥100 points. CDAI is a scoring system for the assessment of Crohn's Disease Activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Time Frame: Baseline and Week 26
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 60.4 [50.2 to 70.0]

11. Secondary Outcome: Part B: Percentage of Participants Achieving Clinical Response at Week 52
Description: as for outcome 10
Time Frame: Baseline and Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 56
percentage of participants | 58.9 [45.0 to 71.9]

12. Secondary Outcome: Part A: Percentage of Participants Achieving Clinical Remission at Week 10
Description: Clinical remission is defined as CDAI score of ≤150 points. CDAI is a scoring system for the assessment of Crohn's Disease Activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease.
Time Frame: Week 10
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 35.6 [26.4 to 45.8]

13. Secondary Outcome: Part A: Percentage of Participants Achieving Clinical Remission at Week 26
Description: as for outcome 12
Time Frame: Week 26
Population: FAS included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 101
percentage of participants | 41.6 [31.9 to 51.8]

14. Secondary Outcome: Part B: Percentage of Participants Achieving Clinical Remission at Week 52
Description: as for outcome 12
Time Frame: Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 56
percentage of participants | 50.0 [36.3 to 63.7]

15. Secondary Outcome: Part B: Percentage of Participants With Durable Clinical Remission
Description: Durable clinical remission is defined as clinical remission at both Week 26 and Week 52. Clinical remission is defined as CDAI score of ≤150 points. CDAI is a scoring system for the assessment of Crohn's Disease Activity, index values of 150 and below are associated with quiescent disease; values above that indicate active disease and values above 450 are seen with extremely severe disease. The percentage of participants assessed at Week 52 who had clinical remission at Week 26 of Part A and also had clinical remission at Week 52 is reported.
Time Frame: Weeks 26 and 52
Population: FAS-Extension is the subset of participants in the FAS who were able to be consented for Part B, based on the timing of Amendment 4. FAS included all enrolled participants who received at least 1 dose of study drug. Participants with missing durable clinical remission status are considered as No durable clinical remission.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 56
percentage of participants | 37.5 [24.9 to 51.5]

ADVERSE EVENTS:
Time Frame: First dose of study drug and up to the last dose or early termination plus 18-week follow-up if applicable (Up to 44 Weeks for Part A Treatment and Up to 70 Weeks for Part B Extension)
Description: At each visit adverse events (AEs) and abnormal laboratory findings reported by participant or observed by the investigator were recorded, irrespective of relation to study treatment. Due to the design of the study, the most common (≥ 5%) non-serious AEs were determined separately for each period of the study, Part A and Part B. A result of 0 in a column means that the event did not meet the ≥ 5% threshold for that study period but did meet the threshold for the other study period.
Groups:
- Vedolizumab 300 mg Part A: Part A: Vedolizumab 300 mg, intravenously (IV), once on Day 1 and Weeks 2, 6, 14 and 22.
- Vedolizumab 300 mg Part B: Following Part A, Part B: Vedolizumab 300 mg, intravenously (IV), once at Weeks 30, 38, and 46.
Arm/Group | Vedolizumab 300 mg Part A | Vedolizumab 300 mg Part B
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/56
Serious Adverse Events (participants affected / at risk) | 12/101 | 6/56
Other Adverse Events (participants affected / at risk) | 26/101 | 9/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg Part A (N=101) | Vedolizumab 300 mg Part B (N=56)
Crohn's disease (Gastrointestinal disorders) | 6 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Infected bite (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg Part A (N=101) | Vedolizumab 300 mg Part B (N=56)
Crohn's disease (Gastrointestinal disorders) | 12 | 5
Viral upper respiratory tract infection (Infections and infestations) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Headache (Nervous system disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT02425111/SAP_000.pdf
  • Study Protocol (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT02425111/Prot_001.pdf